CLINICAL TRIAL: NCT00170157
Title: A Phase II Immunotherapeutic Trial: Combination Androgen Ablative Therapy and CTLA-4 Blockade as a Treatment for Advanced Prostate Cancer
Brief Title: Hormone Therapy and Ipilimumab in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC0253; NCI-2009-01214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0253 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-01

CONDITIONS: Prostate Adenocarcinoma; Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Goserelin; Ipilimumab; CTLA-4 Antigen; Leuprolide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive either leuprolide acetate intramuscularly (IM) or goserelin subcutaneously (SC) on days 0, 28, and 56. Patients also receive oral flutamide three times daily or oral bicalutamide once daily. Treatment with antiandrogen (AA) therapy continues for 3 months (3-4 months for patients who initiated AA therapy <= 21 days prior to enrollment) in the absence of disease progression or unacceptable toxicity. Patients receive ipilimumab IV over 90 minutes on day 7 (within 7-28 days post-initiation of AA therapy for patients who initiated AA therapy <= 21 days prior to enrollment) of AA therapy.
  Interventions: Drug: Bicalutamide; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Ipilimumab; Drug: Leuprolide Acetate; Other: Pharmacological Study
- Arm II (Active Comparator): Patients receive AA therapy as in arm I. Patients may crossover to arm II in the case of disease progression.
  Interventions: Drug: Bicalutamide; Drug: Flutamide; Drug: Leuprolide Acetate; Other: Pharmacological Study

INTERVENTIONS:
Drug: Bicalutamide — Given orally
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Flutamide — Given orally
  Other Names: 4'-Nitro-3'-trifluoromethylisobutyranilide; Apimid; Chimax; Drogenil; Euflex; Eulexin; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolid; Oncosal; Profamid; Prostacur; Prostadirex; Prostica; Prostogenat; SCH 13521; Tafenil; Tecnoflut; Testotard
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
  Arms: Arm I
Drug: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm I
Drug: Leuprolide Acetate — Given IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Other: Pharmacological Study — Correlative study

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide acetate, goserelin, flutamide, or bicalutamide may lessen the amount of androgens made by the body. Monoclonal antibodies, such as ipilimumab, can block cancer growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Giving antihormone therapy together with ipilimumab may kill more tumor cells.

PURPOSE: This randomized phase II trial is study how well giving hormone therapy and ipilimumab together works in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To generally test whether the addition of CTLA-4 blockade can enhance clinical treatment response in advance prostate cancer patients compared with treatment with AA therapy alone.

II. To specifically examine whether concomitant AA therapy + MDX-010 can be used to prolong the progression-free interval in advanced prostate cancer patients compared with inductive short-term AA therapy alone.

III. To specifically examine whether concomitant AA therapy + MDX-010 can be used to enhance initial PSA responses in advanced prostate cancer patients compared with inductive short-term AA therapy alone.

IV. To specifically examine whether delayed MDX-010 can be used to induce PSA response in patients experiencing disease progression following cessation of short-term AA therapy.

V. To generally examine whether MDX-010 enhances host immune response that might be involved in conferring treatment advantages to patients receiving AA therapy.

VI. To specifically examine whether MDX-010 potentiates T-cell responses in advanced prostate cancer patients initiating inductive short-term AA therapy.

VII. To further examine whether treatment induced T-cell responses correlate with clinical response to treatment.

VIII. To examine whether short-term AA there (+/- MDX-010) induces the appearance of newly emigrated T or immature and/or B cells.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive either leuprolide acetate intramuscularly (IM) or goserelin subcutaneously (SC) on days 0, 28, and 56. Patients also receive oral flutamide three times daily or oral bicalutamide once daily. Treatment with antiandrogen (AA) therapy continues for 3 months (3-4 months for patients who initiated AA therapy <= 21 days prior to enrollment) in the absence of disease progression or unacceptable toxicity. Patients receive ipilimumab IV over 90 minutes on day 7 (within 7-28 days post-initiation of AA therapy for patients who initiated AA therapy <= 21 days prior to enrollment) of AA therapy.

Arm II: Patients receive AA therapy as in arm I. Patients may crossover to arm II in the case of disease progression.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* NOTE: All values must be obtained =< 14 prior to study entry
* Histologically confirmed adenocarcinoma of the prostate staged within 180 days of study enrollment, >cT2cN0/M0 stage with or without metastatic disease, with the exclusion of central nervous system (CNS) metastases; includes post radical prostatectomy patients with a rising PSA
* An initial PSA >= 4.0 ng/mL (Hybritech Assay)
* For those patients who have received hormone therapy =< 21 days, a documented PSA of >= 4.0 prior to initiation of hormone therapy is acceptable.
* For patients who are post radical prostatectomy, a rising PSA is acceptable.
* Adequate organ function defined as: WBC >= 3,000/uL; platelets >= 75,000/uL; total bilirubin =< 1.5 mg/dL; transaminases =< 2.5 x upper limit of normal (ULN); serum creatine =< 2.0 mg/dL or calculated creatinine clearance >= 60 mL/min
* ECOG performance status of 0-2
* Able to understand and sign informed consent

Exclusion Criteria:

* Underlying other serious medical condition which, in the opinion of the investigator precludes study participation; this includes immune-suppressive disease such as AIDS or autoimmune disorders such as multiple sclerosis, lupus, or myasthenia gravis
* Patients not recovered from major infections and/or surgical procedures
* Prior hormonal therapy > 21 days prior to enrollment, including estrogens, LH/RH agonists, or antiandrogens
* Recent (=< 3 months of informed consent) usage of immune-suppressive medication including steroids, Immuran, Cyclosporin; topical or inhalational steroid use is permissible
* Prior systemic chemotherapy
* Prior radiation therapy to the prostate
* Prior malignancy, unless the patient has been cancer-free for five years or more
* Uncontrolled underlying medical or psychiatric illness, or serious active infections
* Patient unwilling to complete all required follow-up visits
* History of motor neuropathy considered of the autoimmune origin (e.g. Guillian-Barre Syndrome)
* Concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer
* For patients who elect to undergo the baseline transrectal needle biopsy of the prostate, current usage of systemic anticoagulation therapy, i.e. heparin or Coumadin or inability to discontinue aspirin, aspirin-containing products or ibuprofen for seven days prior to the prostate biopsies required for this study
* No other investigational drugs will be allowed during the study
* Other chemotherapy, radiation therapy, immunotherapy, hormonal therapy, or biologic therapy may not be used while the patient is on study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-06; Primary Completion 2011-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kwon, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 112 participants were recruited between June 2004 and June 2009 at Mayo Clinic.
Pre-assignment Details: All participants were initially randomized to either arm.
Groups:
- Androgen Ablative (AA) Therapy + MDX-010: 3 months of concurrent androgen ablative (AA) therapy + MDX-010
  Androgen ablative (AA) therapy is received a combined regimen of GnRH agonist and androgen receptor blocker. GnRH agonists must be in the form of a 1 month depot of either leuprolide acetate (Lupron) 7.5 mg intramuscular (IM), or goserelin acetate (Zoladex) 3.6 mg subcutaneous (SC) and will be administered on Day 0 (baseline), Day 28 and Day 56. Androgen receptor blockade may be provided by oral administration of either flutamide (Eulexin) 250 mg orally 3 times daily, or bicalutamide (Casodex) 50 mg orally once daily.
  MDX-010 is received as an infusion at a dose of 3.0 mg/kg on day 7.
- Androgen Ablative (AA) Then AA Therapy + MDX-010: 3 months of initial AA therapy alone
  Androgen ablative (AA) therapy is received a combined regimen of GnRH agonist and androgen receptor blocker. GnRH agonists must be in the form of a 1 month depot of either leuprolide acetate (Lupron) 7.5 mg intramuscular (IM), or goserelin acetate (Zoladex) 3.6 mg subcutaneous (SC) and will be administered on Day 0 (baseline), Day 28 and Day 56. Androgen receptor blockade may be provided by oral administration of either flutamide (Eulexin) 250 mg orally 3 times daily, or bicalutamide (Casodex) 50 mg orally once daily.
Period: Treatment Period 1 Initial Randomization
Arm/Group | Androgen Ablative (AA) Therapy + MDX-010 | Androgen Ablative (AA) Then AA Therapy + MDX-010
Started | 54 | 58
Completed | 54 | 58
Not Completed | 0 | 0
Period: Washout Period of 14 Days
Arm/Group | Androgen Ablative (AA) Therapy + MDX-010 | Androgen Ablative (AA) Then AA Therapy + MDX-010
Started | 0 (Participants initially randomized to this arm were not eligible for crossover.) | 58
Completed | 0 | 41
Not Completed | 0 | 17
Period: Treatment Period 2 Crossover
Arm/Group | Androgen Ablative (AA) Therapy + MDX-010 | Androgen Ablative (AA) Then AA Therapy + MDX-010
Started | 0 (Participants initially randomized to this arm were not eligible for crossover.) | 41
Completed | 0 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants initially randomized.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 112
Age, Customized [Number; unit: participants]
  <= 39 | 0
  40-49 | 5
  50-59 | 29
  60-69 | 48
  >= 70 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 112
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Progression-free at 18 Months
Description: PSA progression is defined as a rise in PSA to >4.0 ng/mL demonstrated twice in measurements taken two weeks apart.
Time Frame: 18 months from the start of AA therapy
Measure: Number; unit: participants
Groups:
- Entire Study Population: All participants (Androgen ablative (AA) therapy + MDX-010 and Androgen ablative (AA) therapy alone) initially randomized (i.e., before cross-over) were grouped together for this outcome.
  .
Arm/Group | Entire Study Population
Number analyzed (Participants) | 112
participants | 0

2. Secondary Outcome: Percent of Participants With Undetectable Prostate-specific Antigen (PSA) Response
Description: Percent of participants who had undetectable PSA at 3 months on the initially assigned treatment arm (prior to crossing over).
Time Frame: 3 months
Population: 105 participants had follow-up PSA information; those without a follow-up PSA were excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Androgen Ablative (AA) Therapy + MDX-010 | Androgen Ablative (AA) Then AA Therapy + MDX-010
Number analyzed (Participants) | 53 | 52
percentage of participants | 55 | 39

ADVERSE EVENTS:
Description: Two participants cancelled prior to beginning study treatment, thus did not experience any adverse events.
Groups:
- Entire Study Population: All participants (Androgen ablative (AA) therapy + MDX-010 and Androgen ablative (AA) therapy alone the AA Therapy + MDX-010) were grouped together for this outcome.
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 10/110
Other Adverse Events (participants affected / at risk) | 107/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=110)
Ischemia/Infarction (Cardiac disorders) | 2 (2)
Vision-Blurred (Eye disorders) | 1 (1)
Diarrhea-No Colostom (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Pain-Abdominal (Gastrointestinal disorders) | 1 (1)
Hepatic (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Amylase (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=110)
Anemia (Blood and lymphatic system disorders) | 21 (34)
Lymph node pain (Blood and lymphatic system disorders) | 1 (2)
Cardiovascular (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Endocrine (Endocrine disorders) | 4 (5)
Vision (Eye disorders) | 1 (1)
Vision-Blurred (Eye disorders) | 24 (44)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 2 (2)
Diarrhea-No Colostom (Gastrointestinal disorders) | 8 (8)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Pain-Abdominal (Gastrointestinal disorders) | 1 (1)
Constitutional Symptoms (General disorders) | 5 (5)
Edema: Limb (General disorders) | 3 (4)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 79 (160)
Pain-Chest (General disorders) | 1 (1)
Rigors (General disorders) | 2 (2)
Hepatic (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Abdominal infection (Infections and infestations) | 1 (1)
Colon infection (Infections and infestations) | 1 (1)
Lung (pneumonia) infection (Infections and infestations) | 2 (2)
Penis infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin (cellulites) infection (Infections and infestations) | 1 (2)
Wound infection (Infections and infestations) | 1 (1)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 32 (65)
Alkaline phosphatase (Investigations) | 28 (69)
Amylase (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 31 (55)
Blood bilirubin increased (Investigations) | 22 (36)
Coagulation (Investigations) | 1 (1)
Creatinine (Investigations) | 14 (29)
Lipase increased (Investigations) | 1 (1)
Metabolic/Lab (Investigations) | 10 (12)
Platelet count decreased (Investigations) | 1 (3)
Weight loss (Investigations) | 10 (10)
Bicarbonate (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 24 (37)
Hyperglycemia (Metabolism and nutrition disorders) | 87 (279)
Hyperkalemia (Metabolism and nutrition disorders) | 22 (31)
Hyperuricemia (Metabolism and nutrition disorders) | 18 (34)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 28 (61)
Extremity-lower necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 1 (2)
Ischemia-Cerebral (Nervous system disorders) | 1 (1)
Neuro (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 33 (74)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (3)
Pollakiuria (Renal and urinary disorders) | 75 (171)
Ureteral Obstruction (Renal and urinary disorders) | 1 (1)
Urinary bladder hemorrhage (Renal and urinary disorders) | 10 (11)
Urinary retention (Renal and urinary disorders) | 24 (42)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Prostatic pain (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Nail Changes (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 21 (29)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 88 (207)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes